CLINICAL TRIAL: NCT02171195
Title: A Single Centre, Phase I, Double-blind, Randomised, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetic Profile and Effects on EEG of Single Rising Oral Doses of BIA 2-093 When Given to Healthy Male Adult Volunteers.
Brief Title: A Single Centre, Phase I, Double-blind, Randomised, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetic Profile and Effects on EEG of Single Rising Oral Doses of BIA 2-093
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-2093-101
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Epilepsy
Keywords: Eslicarbazepine acetate; BIA 2-093; Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Group 1 (20 mg) (Experimental)
  Interventions: Drug: BIA 2-093; Drug: Placebo
- Group 2 (50 mg) (Experimental)
  Interventions: Drug: BIA 2-093; Drug: Placebo
- Group 3 (100 mg) (Experimental)
  Interventions: Drug: BIA 2-093; Drug: Placebo
- Group 4 (200 mg) (Experimental)
  Interventions: Drug: BIA 2-093; Drug: Placebo
- Group 5 (400 mg) (Experimental)
  Interventions: Drug: BIA 2-093; Drug: Placebo
- Group 6 (600 mg) (Experimental)
  Interventions: Drug: BIA 2-093; Drug: Placebo
- Group 7 (900 mg) (Experimental)
  Interventions: Drug: BIA 2-093; Drug: Placebo
- Group 8 (1200 mg) (Experimental)
  Interventions: Drug: BIA 2-093; Drug: Placebo

INTERVENTIONS:
Drug: BIA 2-093 — BIA 2-093 20mg, 50 mg, 100 mg, 200 mg, 400 mg, 600 mg, 900 mg, 1200 mg
  Other Names: ESL, Eslicarbazepine acetate
Drug: Placebo — Identical placebo administered as oral tablets with 200 ml potable water.
  Other Names: PLC

SUMMARY:
The purpose of this study is to determine the safety and tolerability of single rising oral doses of BIA 2-093 (proposed doses 20mg, 50mg, 100mg, 200mg, 400mg, 600mg, 900mg and 1200mg) in groups of 8 healthy male adult volunteers.

DETAILED DESCRIPTION:
Single centre, Phase I, double-blind, randomised, placebo-controlled study to investigate single rising oral doses of BIA 2-093 up to 1200 mg in sequential groups of eight healthy male adult subjects. Within each group of eight subjects two subjects were randomised to receive placebo and the remaining six subjects were randomised to receive BIA 2-093. No subject was a member of more than one treatment group. Doses of 20mg, 50mg, 100mg, 200mg, 400mg, 600mg, 900mg and 1200mg were investigated in ascending order. Progression to each dose occurred only after the previous dose level was deemed to be safe and well tolerated by the investigator and the sponsor.

ELIGIBILITY:
Inclusion Criteria:

Adult males aged 18-35 years, with a body mass index (BMI) of 19-28 kg/m2.

* Subjects who were healthy as determined by pre-study medical history, physical examination, 12-lead ECG and EEG.
* Subjects who had clinical laboratory tests acceptable to the investigator.
* Subjects who were negative for HbsAg, anti-HCV and HIV I and II tests at screening.
* Subjects who were negative for drugs of abuse and alcohol tests at screening and admission.
* Subjects who were non-smokers or who smoked less than 10 cigarettes (or equivalent) per day.
* Subjects who were able and willing to give written informed consent.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria.
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity (carbamazepine and related compounds)
* Subjects who had a history of alcoholism.
* Subjects who had a history of drug abuse.
* Subjects who consumed more than 28 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening and/or admission
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or admission (e.g. nausea, vomiting, diarrhoea, heartburn).
* Subjects who had an acute infection such as influenza at the time of screening and/or admission.
* Subjects who had used prescription drugs within 4 weeks of dosing.
* Subjects who had used over the counter medication, excluding routine vitamins but including mega dose vitamin therapy, within one week of dosing.
* Subjects who had used any investigational drug and/or participated in any clinical trial within 3 months of admission to this study.
* Subjects who had donated and/or received any blood or blood products within 3 months prior to screening.
* Subjects who were vegetarians, vegans and/or had medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2000-07; Primary Completion 2000-10 (Actual); Study Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's Drug Research Unit, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo, PLC
- Group 1 20 mg: BIA 2-093 20mg or placebo.
- Group 2 50 mg: BIA 2-093 50mg or placebo
- Group 3 100 mg: BIA 2-093 100mg or placebo
- Group 4 200 mg: BIA 2-093 200mg or placebo
- Group 5 400 mg: BIA 2-093 or 400mg or placebo
- Group 6 600 mg: BIA 2-093 600mg or placebo
- Group 7 900 mg: BIA 2-093 900mg or placebo
- Group 8 1200 mg: BIA 2-093 1200mg or placebo
Period: Overall Study
Arm/Group | Placebo | Group 1 20 mg | Group 2 50 mg | Group 3 100 mg | Group 4 200 mg | Group 5 400 mg | Group 6 600 mg | Group 7 900 mg | Group 8 1200 mg
Started | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Group 1 20 mg | Group 2 50 mg | Group 3 100 mg | Group 4 200 mg | Group 5 400 mg | Group 6 600 mg | Group 7 900 mg | Group 8 1200 mg | Total
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 64
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 64

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Adverse Events
Description: An adverse event was defined as any undesirable event occurring to a subject during the study, whether or not related to the investigational product
Time Frame: up to 20 weeks
Measure: Number; unit: Number of Adverse Events
Arm/Group | Placebo | Group 1 20 mg | Group 2 50 mg | Group 3 100 mg | Group 4 200 mg | Group 5 400 mg | Group 6 600 mg | Group 7 900 mg | Group 8 1200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Number of Adverse Events
  All Adverse Events | 7 | 7 | 3 | 7 | 2 | 1 | 1 | 2 | 7
  AE Considered Not Related to Treatment | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  AE Considered Possibly Related to Treatment | 7 | 5 | 3 | 7 | 2 | 1 | 1 | 2 | 3
  AE of Mild Severity | 7 | 5 | 3 | 6 | 2 | 1 | 1 | 2 | 7
  AE of Moderate Severity | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Group 1 20 mg | Group 2 50 mg | Group 3 100 mg | Group 4 200 mg | Group 5 400 mg | Group 6 600 mg | Group 7 900 mg | Group 8 1200 mg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/16 | 4/6 | 2/6 | 3/6 | 2/6 | 1/6 | 1/6 | 1/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Group 1 20 mg (N=6) | Group 2 50 mg (N=6) | Group 3 100 mg (N=6) | Group 4 200 mg (N=6) | Group 5 400 mg (N=6) | Group 6 600 mg (N=6) | Group 7 900 mg (N=6) | Group 8 1200 mg (N=6)
Mouth dry (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 2 | 2 | 2 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Psychiatric disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper resp tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other